CLINICAL TRIAL: NCT03179735
Title: Mouthwashes as Positive Modulators of Periodontal Response During Orthodontic Treatment: a 6-month Randomized Placebo Controlled Clinical Trial
Brief Title: Mouthwashes During Orthodontic Treatment
Acronym: MOUORT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Taubate (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MOUORT
Record Dates: First submitted 2017-06-01; First posted 2017-06-07 (Actual); Last update posted 2017-06-07 (Actual); Status verified 2017-06

CONDITIONS: Gingivitis
MeSH Terms: conditions — Gingivitis | interventions — Oils, Volatile; Cetylpyridinium

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Essential oils mouthwash (Experimental): Essential-oils group will rinse with an alcohol-free mouthwash (twice daily use; 20 ml/30 s) containing a fixed combination of four essential oils (eucalyptol 0.092%, menthol 0.042%, methyl salicylate 0.060%, thymol 0.064%)
  Interventions: Drug: Essential oils
- Cetylpyridinium mouthwash (Experimental): Cetylpyridinium chloride group will rinse with an alcohol-free mouthwash (twice daily use; 20 ml/30 s) containing cetylpyridinium chloride 0.7 mg/ml
  Interventions: Drug: Cetylpyridinium Chloride 0.7 mg/ml
- Placebos mouthwash (Placebo Comparator): Placebo group will rinse with an alcohol-free placebo solution (twice daily use; 20 ml/30 s)
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Essential oils — Patients will be submitted to one-stage ultrasonic debridement to remove plaque, stain(s), and any possible supragingival dental calculus. Further, oral instructions and an oral hygiene kit with fluoride dentifrice, toothbrush and plastic cups marked to indicate the rinse volume will be provided. According to study group, the first rinse will be performed under supervision at the study center and the remaining rinses will be performed unsupervised at home.
  First rinse will be performed 15 days before orthodontic appliances bonding while the last rinse will be performed 6 months after bonding.
  Arms: Essential oils mouthwash
Drug: Cetylpyridinium Chloride 0.7 mg/ml — Patients will be submitted to one-stage ultrasonic debridement to remove plaque, stain(s), and any possible supragingival dental calculus. Further, oral instructions and an oral hygiene kit with fluoride dentifrice, toothbrush and plastic cups marked to indicate the rinse volume will be provided. According to study group, the first rinse will be performed under supervision at the study center and the remaining rinses will be performed unsupervised at home.
  First rinse will be performed 15 days before orthodontic appliances bonding while the last rinse will be performed 6 months after bonding.
  Arms: Cetylpyridinium mouthwash
Drug: Placebos — Patients will be submitted to one-stage ultrasonic debridement to remove plaque, stain(s), and any possible supragingival dental calculus. Further, oral instructions and an oral hygiene kit with fluoride dentifrice, toothbrush and plastic cups marked to indicate the rinse volume will be provided. According to study group, the first rinse will be performed under supervision at the study center and the remaining rinses will be performed unsupervised at home.
  First rinse will be performed 15 days before orthodontic appliances bonding while the last rinse will be performed 6 months after bonding.
  Arms: Placebos mouthwash

SUMMARY:
The number of orthodontic treatment provided to Brazilian population has been increased. Unfortunately, some negative effects such as gum bleeding and bad breath are commonly observed. It partially happens because tooth brushing and flossing become more difficult in the presence of braces. Therefore, there is a need for clinical protocols able to maintain the mouth healthy during orthodontic treatment.

Considering that proper use of mouthwashes by in individuals without braces is accompanied by decrease in plaque and gum inflammation levels, it was hypothesized that, during orthodontic treatment their anti-gingivitis and anti-plaque properties would positively affect oral health. Objectives: The present study will compare the effects of two commercially available mouthwashes with a placebo mouthwash in orthodontic patients wearing fixed appliances.

Whole-mouth clinical examinations will be performed in periodontally healthy patients 15 days before, at the day of bonding and also 3 and 6 months after braces bonding. Hard and soft tissues status, presence of gingivitis and amount of dental plaque will be monitored to determine mouthwashes efficacy. At these same time-points plaque samples will be collected from dental sites and braces surfaces aiming at determining total levels of bacteria and levels of specific bacteria related to gum disease. After a full-mouth ultrasonic debridement to remove dental plaque, stains and tartar, patients will be randomly assigned to an Essential oils, Cetylpyridinium chloride or a placebo mouthwash for 6 months (40 ml/day). Further, samples of orthodontic wires will be analyzed under microscopy to check whether regular use of mouthwashes increases the risk of corrosion or not.

ELIGIBILITY:
Inclusion Criteria:

* good general health;
* class I or class II malocclusions with a nonsurgical orthodontic treatment plan for alignment and leveling including no-extraction, extraction of two upper premolars or extraction of four premolars; no previous orthodontic treatment; overbite and overjet that allowed brackets to be placed on the lower teeth without occlusal interferences;
* periodontal health (with no clinical signals of inflammation, GI <1 e no clinical attachment loss);
* at least 26 natural teeth;

Exclusion Criteria:

* severe skeletal malocclusion in anteroposterior, vertical or transverse dimensions; surgical orthodontic plan;
* mouth breathing;
* gingivitis; periodontitis; gingival overgrowth;
* prosthetic fixed devices, removable partial dentures or overhanging restorations;
* systemic diseases or conditions that could influence the periodontal status;
* smokers and former-smokers;
* pregnancy or breast-feeding;
* history of sensitivity or suspected allergies following the use of oral hygiene products; any antibiotic prophylaxis;
* antibiotics and/or anti-inflammatory drug use in the six months prior to the beginning of the study;
* regular use of chemotherapeutic antiplaque/antigingivitis products;
* periodontal treatment performed within six months prior to study initiation;
* unwillingness to return for follow-up.

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-03-10 (Estimated); Study Completion 2018-07-10 (Estimated)

PRIMARY OUTCOMES:
Changes in gingival index | up to 6 months
  Gingival index changes (mean scores) from baseline to 6 months.

SECONDARY OUTCOMES:
Changes in plaque index | up to 6 months
  Plaque index changes (mean scores) from baseline to 6 months.
Changes in subgingival bacterial levels | up to 6 months
  Changes in bacterial levels (total number of bacterial cells and specific numbers of Actinomyces naeslundii, Streptococcus oralis, Fusobacterium nucleatum, Aggregatibacter actinomycetemcomitans, Porphyromonas gingivalis, Tannerella forsythia, Treponema denticola) from sub gingival samples.
Changes in bracket bacterial levels | up to 6 months
  Changes in bacterial levels (total number of bacterial cells and specific numbers of Actinomyces naeslundii, Streptococcus oralis, Fusobacterium nucleatum, Aggregatibacter actinomycetemcomitans, Porphyromonas gingivalis, Tannerella forsythia, Treponema denticola) from bracket samples.
Changes in gingival overgrowth measurements | up to 6 months
  Gingival overgrowth changes (mean scores) from baseline to 6 months.
Corrosion of orthodontic devices | up to 6 months
  Percentage of areas of orthodontic devices showing corrosive superficial changes at 3 and 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Sheila C Cortelli, PhD, Principal Investigator — Dean periodontics department
Locations (1):
- Nucleus of periodontal research of University of Taubate, Taubaté, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared.